CLINICAL TRIAL: NCT05821517
Title: METHOXYFLURANE or Virtual Reality Headset vs Standard Analgesic Management for the Reduction of Anterior Shoulder Dislocation
Brief Title: METHOXYFLURANE or Virtual Reality Headset vs Standard Analgesic Management for the Reduction of Anterior Shoulder Dislocation (HYPNOLUX)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-AOI-11
Record Dates: First submitted 2023-03-10; First posted 2023-04-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Anterior Shoulder Dislocation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Active Comparator): An anticipated analgesia protocol composed of PARACETAMOL 1g +/- OXYNORM 5 mg or 10 mg according to patients weight and pain intensity as evaluated by a simple numeric rating scale is administred prior to the reduction procedure. Inhaled equimolar mixture of oxygen and notrous oxyde (MEOPA) at a 15L/min flux is administered concomitantly to the reduction procedure.
  Interventions: Drug: Standard of care
- Medical device : VR headset (Experimental): Use of a " virtual reality " (VR) headset of " Pico G2 " type with " HypnoVR " software and audio headset " Taotronics BH22 " during all the reduction care
  Interventions: Device: Helmet virtual reality.
- Medication : Methoxyflurane analgesia (Experimental): Self administered inhalated methoxyflurane (maximal inhaled dose : 3 mL)
  Interventions: Drug: Administration of METHOXYFLURANE

INTERVENTIONS:
Device: Helmet virtual reality. — Use of a " virtual reality " (VR) headset of " Pico G2 " type with " HypnoVR " software and audio headset " Taotronics BH22 " during all the reduction care
  Arms: Medical device : VR headset
Drug: Administration of METHOXYFLURANE — Self administered inhalated methoxyflurane (maximal inhaled dose : 3 mL)
  Arms: Medication : Methoxyflurane analgesia
Drug: Standard of care — An anticipated analgesia protocol composed of PARACETAMOL 1g +/- OXYNORM 5 mg or 10 mg according to patients weight and pain intensity as evaluated by a simple numeric rating scale is administred prior to the reduction procedure. Inhaled equimolar mixture of oxygen and notrous oxyde (MEOPA) at a 15L/min flux is administered concomitantly to the reduction procedure.
  Arms: Standard of care

SUMMARY:
Anterior shoulder dislocation is a pathology frequently encountered in emergency medicine.

The success in reducing anterior shoulder dislocations depends on muscle relaxation, which is itself conditioned by the patient's pain and apprehension. However, there is no consensus on the optimal technique for reducing anterior shoulder dislocation or the analgesia associated with it.

Analgesia with METHOXYFLURANE showed a greater reduction in post-traumatic pain compared to standard analgesic treatment and faster action of METHOXYFLURANE. A retrospective study which has compared analgesia with METHOXYFLURANE and analgesic sedation with PROPOFOL found a shoulder reduction success rate of 80% and a reduction in the average length of stay in the emergency department.

Finally, the use of virtual reality in pain management is emerging in our practices by allowing pre- and per-procedure hypno-sedation-analgesia. However, the use of virtual reality headsets has not been studied in the management of anterior shoulder dislocation.

The use of these two techniques could therefore limit the use of procedural sedation in the context of shoulder dislocation reduction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and/or breastfeeding women and women of childbearing age who do not have effective contraception (hormonal, mechanical or surgical).
* Patients with difficulties in understanding or using the devices studied.
* Patients with a contraindication to the use of one of the studied devices.
* Patients with a history of relevant shoulder surgery
* Presence of other associated trauma,
* Previous inclusion in the same study

Exclusion Criteria:

* Withdrawal of voluntary informed consent from the patient
* Violation of protocol
* Presence of a fracture associated with the dislocation (excluding Malgaigne's notches)
* Posterior, inferior or erecta dislocation
* Presence of initial vascular and nerve complications
* Any indication for surgical management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Decrease in the rate of procedural sedation of anterior shoulder dislocation | Day 1 (day of reduction of anterior shoulder dislocation)
  Rate of use of procedural sedation for anterior shoulder dislocation reduction in the interventional groups compared to the control group

SECONDARY OUTCOMES:
The amount of co-antalgesics administered | 3 months
  Posology of co-analgesic medications administered
The duration of the procedure | Day 1 (day of change of anterior shoulder dislocation)
  Time lenght of the reduction procedure
The dosage of drugs used in procedural sedation | Day 1 (day of reduction of anterior shoulder dislocation)
  Posology of sedative drugs administered for a procedural sedation
The average length of stay in the emergency department | 3 months
  Average length of stay in the emergency department
Patient satisfaction | 3 months
  Patient satisfaction at the end of care evaluated with a questionnaire EVA
The rate of reduction-related complications | 3 months
  Complications related to the reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No